CLINICAL TRIAL: NCT06168864
Title: Development of Artificial Intelligence Models for Segmentation and Characterization of Prostate Cancer: a Single-center Retrospective Observational Study.
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: AI_Pca
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Artificial intelligence models for segmentation and characterization of prostate cancer — rtificial intelligence algorithms for the automatic segmentation of prostate cancer lesions on medical images.

SUMMARY:
Prostate cancer is the second most common cancer in the male population. This pathology represents an oncological and public health problem especially in developed countries, due to a greater presence of elderly men in the population.

Medical imaging plays a central role in the staging and restaging of prostate disease. Magnetic resonance imaging (MRI), computed tomography (CT) and positron emission tomography (PET) are among the methods commonly used in normal clinical practice for the characterization of prostate cancer. To date, the study of these images is limited to a qualitative visual analysis, however there is increasing evidence relating to the usefulness of introducing a quantitative (or semi-quantitative) analysis of biomedical images.

The current increase in available imaging data, and their quality, allows the application of artificial intelligence methods also in the medical field for the automation of tasks (e.g. automatic segmentation) and classification (e.g. tumor aggressiveness).

The extraction of quantitative data, and more generally the study of tumor lesions, requires manual segmentation by one or more doctors. This process requires very long times as each image must be processed individually; furthermore, the result also depends on the level of experience of the doctor carrying out the segmentation and this could create a source of heterogeneity, affecting the reproducibility of the segmentation.

AI-based automatic segmentation methods can be applied to medical images for the localization of tumor lesions, thus exceeding the limits of manual segmentation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological diagnosis of prostate cancer;
* Patients who performed a PET exam with 68 Ga-PMSA.

Exclusion Criteria:

* CT and MR images with artifacts that preclude interpretation of results.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer undergoing PET examination with 68 Ga-PMSA (PET/CT or PET/MRI), since 01/06/2020, at the U.O. of Nuclear Medicine at the San Raffaele Hospital on the clinical indication of the specialist.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Artificial intelligence algorithms for the classification of prostate cancer lesions on medical images. | 2 years
  PET images from enrolled patients will be used to create models that investigate the ability of artificial intelligence to automate tumor segmentation tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No